CLINICAL TRIAL: NCT04392817
Title: Formulatin and Application of a Remediation Software Porgram for Correction of Articulatory Errors in Patients With Velopfaryngeal Dysfunction
Brief Title: Efficacy of an Arabic Articulatory Error Remediation Software Program in Patients With Velopharyngeal Valve Dysfunction:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mamdouh (Other)
Responsible Party: Sponsor-Investigator, Alaa Mamdouh, Assistant lecturer of phoniatrics, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0105440
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Velopharyngeal Insufficiency; Articulation Disorders; Hypernasality Syndrome Due to Velopharyngeal Weakness
Keywords: Velopharyngeal dysfunction Hypernasality
MeSH Terms: conditions — Velopharyngeal Insufficiency; Articulation Disorders

STUDY DESIGN:
Intervention Model Description: a quasi experimental study comparing pre to post therapy intervention in one group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the participating group in the intervention (Experimental): patient complaining of seppch rerrors due t ovelopharyngeal insufficiency and underwent the intervention
  Interventions: Behavioral: Arabic Articulatory Error Remediation software program

INTERVENTIONS:
Behavioral: Arabic Articulatory Error Remediation software program — A speech therapy computerized intervention

SUMMARY:
To develop a remediation software program that is specific for correcting speech errors in patients with velopharyngeal dysfunction in the Arabic language and test its efficacy, on one group comparing pre and post results

DETAILED DESCRIPTION:
The study was carried on 40 patients having articulation errors in cases of velopharyngeal valve dysfunction attending the unit of phoniatrics, otorhinolaryngology department, Alexandria University.

The patients met the specified inclusion and exclusion criteria. The patient underwent pre intervention evaluation and 3 parameters were chosen to compare efficacy of the program before and after therapy.

these include auditory perceptual assessment of speech, nasometer test and articulation test.

The patient underwent the remediation software program as individual sessions. then after finishing the therapy, the patients underwent post therapeutic evaluation with the 3 specified criteria

Statistical analysis Was carried out using SPSS statistics software version 23. Quantitative data were tested for normality using the Kolmogorov-Smirnov test. The variables which were normally distributed were described by Mean± SD. The variables which were not normally distributed, were described by median (Min-Max). Qualitative data were expressed by numbers and percentages. The results were calculated at a level of significance of 5% or less.

ELIGIBILITY:
Inclusion Criteria:

* clinically presented by articulation errors due to velopharyngeal dysfunction
* Age of 5 years and above with
* must have normal hearing and vision.

Exclusion Criteria:

* Unrepaired cleft palate.
* Large palatal fistula.
* Brain damage and intellectual disability.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
change in Arabic articulation test | base line( pre -intervention)
  a qualitative test that define presence or absence of articulation errors
change in Arabic articulation test | immediately after intervention
  a qualitative test that define presence or absence of articulation errors
change in naso meter values | pre intervention
  a device that measure nasalance score as a ratio expressed in percentage between nasal sound energy to nasal plus oral sound in patients pre and post intervention for quantitaive assesment of nasal air emission and nasal tone where the lower values mean beteer results
change in naso meter values | immediately after intervention
  a device that measure nasalance score as a ratio expressed in percentage between nasal sound energy to nasal plus oral sound in patients pre and post intervention for quantitaive assesment of nasal air emission and nasal tone where the lower values mean beteer results
change in Auditory perceptual assessment of speech | pre intervention
  A qualitative scale of patient speech : 5 grade from 0( not present) to 4 (sever)
change in Auditory perceptual assessment of speech | immediately after intervention
  A qualitative scale of patient speech : 5 grade from 0( not present) to 4 (sever)

SECONDARY OUTCOMES:
effect of the age factor on nasometer values after intervention | immediately after intervention
  statistical tests for correlation
effect of the age factor on auditory perceptual assessment after intervention | immediately after intervention
  statistical tests for correlation
effect of the surgical repair on the nasometer values after intervention | immediately after intervention
  comparison between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Engy S Elhakeem, PhD, Study Director — Otorhinolaryngology department,Faculty of Medicine, Alexandria University; Reham M Elmaghraby, PhD, Study Chair — Otorhinolaryngology department,Faculty of Medicine, Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria universtiy, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there will be a palne to make IPD available
Supporting Information: Study Protocol, SAP
Time Frame: for 6 months after puplishing
Access Criteria: Through the Email Address A_abdelhamed14@alexmed,edu,eg

REFERENCES:
- [Background] Siegel-Sadewitz VL, Shprintzen RJ. Changes in velopharyngeal valving with age. Int J Pediatr Otorhinolaryngol. 1986 Apr;11(2):171-82. doi: 10.1016/s0165-5876(86)80011-8. PMID 3744698
- [Background] Ha S, Cho SH. Nasalance scores for normal Korean-speaking adults and children: Effects of age, vowel context, and stimulus length. Int J Pediatr Otorhinolaryngol. 2015 Aug;79(8):1235-9. doi: 10.1016/j.ijporl.2015.05.019. Epub 2015 Jun 4. PMID 26089139
- [Background] Phua YS, de Chalain T. Incidence of oronasal fistulae and velopharyngeal insufficiency after cleft palate repair: an audit of 211 children born between 1990 and 2004. Cleft Palate Craniofac J. 2008 Mar;45(2):172-8. doi: 10.1597/06-205.1. PMID 18333650
- [Background] Sell D. Issues in perceptual speech analysis in cleft palate and related disorders: a review. Int J Lang Commun Disord. 2005 Apr-Jun;40(2):103-21. doi: 10.1080/13682820400016522. PMID 16101269
- [Background] Brunnegard K, Lohmander A, van Doorn J. Comparison between perceptual assessments of nasality and nasalance scores. Int J Lang Commun Disord. 2012 Sep-Oct;47(5):556-66. doi: 10.1111/j.1460-6984.2012.00165.x. Epub 2012 Jul 25. PMID 22938066
- [Background] Kummer AW( 2104) Cleft Palat and Craniofacial Anomalies: Effect on speech and resonance, 3rd edition ed. Delmar Cengage, NY. 23-31 p. .
- [Background] Dudas JR, Deleyiannis FW, Ford MD, Jiang S, Losee JE. Diagnosis and treatment of velopharyngeal insufficiency: clinical utility of speech evaluation and videofluoroscopy. Ann Plast Surg. 2006 May;56(5):511-7; discussion 517. doi: 10.1097/01.sap.0000210628.18395.de. PMID 16641626
- [Background] 3. Kirschner RE, Baylis AL(2013) Velopharyngeal dysfunction. In: Neligan PC, Gurtner GC, editors. Plastic Surgery: Principles and practice, 3rd ed. Elsevier Inc, St. Louis. p. 614-30.
- [Background] Kotby MN, Bassiouny S, El-Zomor M, E M, editors.(1986) Standardization of an Articulation Test (In Arabic). Proceeding of the 9th Annual Ain Shams Medical Congress, Cairo, Egypt.
- [Background] Abou-Elsaad T, Baz H, Afsah O, Mansy A. The nature of articulation errors in Egyptian Arabic-speaking children with velopharyngeal insufficiency due to cleft palate. Int J Pediatr Otorhinolaryngol. 2015 Sep;79(9):1527-32. doi: 10.1016/j.ijporl.2015.07.003. Epub 2015 Jul 14. PMID 26209352
- [Background] 18. Kotby MN E-SA, Alloush T, Gamal N(1992) 3. Dysarthria Annual Bulletin of Yufuin Kosenenkin Hospital. Hiese. 373-80.